CLINICAL TRIAL: NCT02206269
Title: Registry of Bronchial Thermoplasty (BT) Procedures in China
Brief Title: China Alair System Registry Study-CARE Study
Acronym: CARE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: BSC International Medical Trading (Shanghai) Co., Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: E7100
Record Dates: First submitted 2014-07-24; First posted 2014-08-01 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alair System: This is a single arm study with Alair system used.
  Interventions: Device: Alair System

INTERVENTIONS:
Device: Alair System — The Alair system is used for doing bronchial thermoplasty.

SUMMARY:
The objective of this Registry is to collect real-world outcome data for bronchial thermoplasty (BT) procedures in patients with severe persistent asthma who remain symptomatic despite taking standard of care maintenance medications.

DETAILED DESCRIPTION:
Data will be used to confirm the impact of BT on safety, effectiveness, quality of life, and the anticipated reduction in healthcare utilization events and cost by way of a reduction in severe asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult aged 18 years or older with severe persistent asthma who remains symptomatic despite taking standard of care maintenance medications.
2. Patient is able to read, understand, and sign a written Informed Consent to participate in the Registry and able to comply with the study requirements.
3. Patient is able to undergo bronchoscopy in the opinion of the Investigator or per hospital guidelines and as described in the Alair System Directions for Use (DFU).

Exclusion Criteria:

1. Patient has an implanted electrical stimulation device (e.g., a pacemaker, cardiac defibrillator, or deep nerve or deep brain stimulator).
2. Patient has any other medical condition that would make them inappropriate for study participation, in the Investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The real world patient polulaiton who undergo BT in China
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe asthma exacerbations following BT with the Alair System. | 1 year
  Severe asthma exacerbation is defined as worsening of asthma symptoms requiring use of systemic corticosteroids (tablets, suspension, or injection) (NAEPP Guidelines, 2007).
  For patients already taking oral corticosteroids on a daily or alternate day basis, a severe asthma exacerbation is defined as a worsening of asthma symptoms requiring any increase in daily dose of systemic corticosteroids.
  For consistency, courses of corticosteroids separated by 1 week or more will be treated as separate severe exacerbations.

SECONDARY OUTCOMES:
Quarlity of life of Patients | 1 year
  Asthma Quality of Life Questionnaire (AQLQ) score Asthma Control Questionnaire(ACQ)
Health care utilization | 1 year
  Emergency Department Visits,Hospitalizations,Unscheduled office visits including urgent care visits
FEV1 | 1 year
  Pre- and post-bronchodilator FEV1
Serious respiratory adverse events | 1 year
  Rates of and proportion of patients with serious respiratory adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Lin, Professor, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- BSC International Medical Trading (Shanghai) Co., Ltd., Shanghai, Shanghai Municipality, China